CLINICAL TRIAL: NCT06633458
Title: Adolescent Psychiatry Inpatients: Self-reported Parent-adolescent Communication Quality As a Predictor of Treatment Outcome
Brief Title: Adolescent Psychiatry Inpatients: Self-reported Parent-adolescent Communication Quality and Treatment Outcome
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: JuStCom
Record Dates: First submitted 2024-07-30; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-07

CONDITIONS: Mental Disorder in Adolescence; Depression in Adolescence; Anxiety
Keywords: mental health; adolescence; communication
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group (observation only): Adolescent inpatients at the child and adolescent psychiatry, age 14-17 years.

SUMMARY:
The quality of parent-adolescent communication has been found to be associated with adolescent mental health. However, little is known about the association of parent-adolescent communication and adolescent mental health in the context of psychiatry inpatient treatment.

This study aims to find out whether self-reported parent-adolescent communication quality at the time of admission to psychiatry predicts the treatment outcome in terms of symptom reduction 6 months later in an adolescent inpatient sample. It also aims to track changes in adolescent self-reported communication quality in the course of inpatient treatment and afterwards (2, 4 and 6 months after admission) to see whether improvement predicts treatment outcome, with treatment outcome being defined as symptom reduction to baseline. As a secondary endpoint, it will be assessed whether a placement of the adolescent outside the family was considered during treatment and whether self-reported communication quality at the time of admission predicts the consideration of placement outside the family.

DETAILED DESCRIPTION:
The main hypotheses of the study are:

1a Higher quality of self-reported parent-adolescent communication at baseline is positively associated with higher symptom reduction from baseline (psychiatry admission, t0) to 6 months after admission (t3).

1. b Higher improvement of parent-adolescent communication from t0 to t3 is positively associated with higher symptom reduction from t0 to t3.
2. Higher quality of self-reported parent-adolescent communication at baseline is negatively associated with consideration of the adolescent's placement outside the family during treatment.

The hypotheses 1a and 1b will be assessed with a linear regression model, hypothesis 2 will be assessed with a logistic regression model.

Covariates that will be taken into consideration are symptom severity at baseline, socioeconomic status of the family, adolescent gender, age, and comorbidity. Sensitivity analyses will be calculated for inpatient treatment duration and outpatient treatment duration after discharge from the hospital.

Symptom severity as the primary outcome is assessed with three measures: YSR (Youth Self-Report), DISYPS-ANG (Diagnostik-System für Psychische Störungen - Angststörungen) and DISYPS-DES Diagnostik-System für Psychische Störungen - Depressive Störungen). The relevant scale will be chosen according to the primary clinical diagnosis: If the primary diagnosis is anxiety (F40-F41), DISYPS-ANG will be used for the primary outcome. If the primary diagnosis is depression (F32-F33), DISYPS-DES will be used. If any other condition is the primary diagnosis, the YSR total scale will be used. Raw values of the DISYPS and the YSR will be transformed into z-values.

ELIGIBILITY:
Inclusion Criteria:

* Admission to inpatient care unit of the adolescent psychiatry at the University Medical Center Hamburg-Eppendorf.

Exclusion Criteria:

* Severe symptom burden at admission
* Lack of knowledge of the German language.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents aged 14;1 to 17;12 years with a diagnosis of a mental disorder requiring inpatient treatment at a psychiatric site.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-07-07 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in self-rated relevant symptoms according to the discharge diagnosis (general mental health) | From baseline to 6 months after admission (T3)
  General mental health symptoms will be assessed with the YSR (Youth Self-Report). If a condition other than F32-33 or F40-41 is the primary diagnosis, the YSR total scale will be used. The YSR consists of 112 items, rated on a three-step scale. Higher values indicate higher symptom burden.
Change in self-rated relevant symptoms according to the discharge diagnosis (depression symptoms) | From baseline to 6 months after admission (T3)
  Depression symptoms will be assessed with the DISYPS-DES (Diagnostik-System für Psychische Störungen - Depressive Störungen). If the primary diagnosis is depression (F32-F33), DISYPS-DES will be used. The DISYPS-DES consists of consist of 29 items, rated on a four-step scale. Higher values indicate higher symptom burden.
Change in self-rated relevant symptoms according to the discharge diagnosis (anxiety symptoms) | From baseline to 6 months after admission (T3)
  Anxiety symptoms will be assessed with the DISYPS-ANG (Diagnostik-System für Psychische Störungen - Angststörungen). If the primary diagnosis is anxiety (F40-F41), DISYPS-ANG will be used for the primary outcome. The DISYPS-ANG consists of 44 items, rated on a four-step scale. Higher values indicate higher symptom burden.
Discussion of external placement (rated by clinician) | From baseline to 6 months after admission (T3)
  The responsible clinician rates whether an external placement (outside the family) of the adolescent was discussed in the context of psychiatric treatment (yes/no). It has to be considered as discussed ("yes") if either the adolescent, one parent or more or the treatment team articulate a wish/recommendation regarding external placement during the period of treatment toward any other party.

SECONDARY OUTCOMES:
Change in self-rated parent-adolescent communication quality | From baseline to 6 months after admission (T3)
  PACS (Parent-Adolescent Communication Scale) questionnaire. The PACS consists of 20 items rated on a five-step scale and ranges from 20-100 with better values indicating higher communication quality.

CONTACTS AND LOCATIONS:
Overall Officials: Holger Zapf, Dr, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided